CLINICAL TRIAL: NCT04988542
Title: Clinical Efficacy of a Novel Delivery Supplement on Sleep Quality
Brief Title: Clinical Efficacy of a Supplement on Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TruDiagnostic (Industry)
Collaborators: Circadian Wellness Corp (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TD-SQ-001
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Patients will be in the control group for 1 month and in the intervention group for one month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep supplement (Experimental): Circadian Wellness sleep SL strip nightly for 30 days.
  Interventions: Dietary Supplement: Circadian Wellness sleep SL strip
- Control Group (Placebo Comparator): Participants in the control group will have no intervention and no change in their usual daily routine or supplements. They will be asked to not take any sleep aid supplement during the study period.
  Interventions: Dietary Supplement: Circadian Wellness sleep SL strip

INTERVENTIONS:
Dietary Supplement: Circadian Wellness sleep SL strip — Participants in the intervention group will be asked to begin Circadian Wellness sleep SL strip nightly for 30 days. Participants will continue the supplementation for the 30 days.

SUMMARY:
This is a prospective randomized clinical study of 30 patients to evaluate a novel sleep supplement. This study will be evaluating the effectiveness of the supplement over a 2 month program. The study will assess the effects that the supplement has on a patient's sleep metrics and epigenetic age biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of any ethnicity.
* Age Range - 16 - 65
* Patient must be able to comply with treatment plan and laboratory tests

Exclusion Criteria:

* Neoplastic cancer within 5 years prior to screening, except for cutaneous basal cell or squamous cell cancer resolved by excision
* No immune system issues or immunodeficiency disease
* No history of viral illness which could be reactivated by immune downregulation
* Presence of clinically significant acute or unstable cardiovascular and cerebrovascular (stroke)
* Diagnosis of a transient ischemic attack in the 6 months prior to screening
* Patients infected with hepatitis, C or HIV
* Patients with Body Mass Index (BMI) > 40 kg/m2
* Presence of active infection
* Any other illness, psychiatric disorder, alcohol or chemical dependence that in the opinion of the investigator would render a patient unsuitable to participate in the study
* Unable or unwilling to provide required blood sample for testing
* As for the male-participants they are recommended to avoid fertilization for the first 6 months after the clinical trial.
* If the patient has previously used any products in a month prior to the start of the trial.
* Known sleep disorder ie. obstructive sleep apnea
* Presence of schizophrenia, bipolar disorder
* Concurrent use of cannabis

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-30 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Epigenetic Age | Change from baseline to 2 months

SECONDARY OUTCOMES:
Sleep duration | change from baseline to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Goel, Principal Investigator — Peak Human Labs

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cui XY, Cui SY, Zhang J, Wang ZJ, Yu B, Sheng ZF, Zhang XQ, Zhang YH. Extract of Ganoderma lucidum prolongs sleep time in rats. J Ethnopharmacol. 2012 Feb 15;139(3):796-800. doi: 10.1016/j.jep.2011.12.020. Epub 2011 Dec 21. PMID 22207209